CLINICAL TRIAL: NCT04157543
Title: Single-blinded, Randomized Preliminary Study Evaluating the Effects of Electroacupuncture for Postoperative Pain Relief in Patients With Arthroscopic Repair for Triangular Fibrocartilage Complex (TFCC) Tears
Brief Title: A Study Evaluates the Effects of Electroacupuncture for Postoperative Pain Relief in Patients With Repair for TFCC Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH108-REC1-035
Record Dates: First submitted 2019-04-22; First posted 2019-11-08 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain Relief
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture (Experimental): electroacupuncture at points after surgery
  Interventions: Other: electroacupuncture
- electroacupuncture non-point (Sham Comparator): electroacupuncture at non-points after surgery
  Interventions: Other: electroacupuncture
- Control group (No Intervention): only injection painkiller were used before surgery

INTERVENTIONS:
Other: electroacupuncture — acupuncture with electricity
  Arms: electroacupuncture; electroacupuncture non-point

SUMMARY:
Triangular Fibrocartilage Complex (TFCC) is the main stable structure of the distal ulnar joint (DRUJ), and the damage of the triangular fibrocartilage complex is the most common cause of pain in the ulnar side of the wrist in the young athlete population. Once TFCC is injured, arthroscopic surgery is a common repair method. The postoperative analgesic method is generally oral or injection analgesic. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. However, there is no evaluation of analgesic efficacy after arthroscopic repair of the TFCC. Therefore, it is hoped that the efficacy of electroacupuncture for analgesia after arthroscopic repair of the TFCC is demonstrated by this study. And, the investigators also hope the investigators can reduce the use of painkillers through electroacupuncture.

Methods:It is expected that 30 patients will be randomly assigned to the following groups: electroacupuncture group(EAG), EA at points; non-point group (NPG), EA at non-points, control group (CG) without EA

1. electroacupuncture group(EAG): EA at points after surgery
2. non-point group (NPG): EA at non-points after surgery
3. Control group: only injection painkiller were used before surgery

DETAILED DESCRIPTION:
Triangular Fibrocartilage Complex (TFCC) is the main stable structure of the distal ulnar joint (DRUJ), and the damage of the triangular fibrocartilage complex is the most common cause of pain in the ulnar side of the wrist in the young athlete population. Once TFCC is injured, arthroscopic surgery is a common repair method. The postoperative analgesic method is generally oral or injection analgesic. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. However, there is no evaluation of analgesic efficacy after arthroscopic repair of the TFCC. Therefore, it is hoped that the efficacy of electroacupuncture for analgesia after arthroscopic repair of the TFCC is demonstrated by this study. And, the investigators also hope the investigators can reduce the use of painkillers through electroacupuncture.

Methods:

It is expected that 30 patients will be randomly assigned to the following groups: electroacupuncture group(EAG), EA at points; non-point group (NPG), EA at non-points, control group (CG) without EA

1. electroacupuncture group(EAG): EA at points after surgery
2. non-point group (NPG): EA at non-points after surgery

Mode of operation: After the patient has returned to the recovery room, take the needle after 30 minutes, and then statistics.

Acupoint selection:

1. true acupoints: needles were inserted to Kunlun(BL60) and Sanyinjiao(SP6) contralateral to the operated leg and deqi sensation elicited at acupoints
2. false point: the needles were inserted to Zusanli(ST36) and Shangjuxu(ST37) contralateral to the operated leg and deqi sensation elicited at acupoints
3. Control group:only injection and oral painkiller were used before surgery

Data collection:

1. Record the time required for the first injection of analgesics
2. The number of doses of injection painkiller used in 36 hours after surgery (count)

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic specialist diagnoses tearing of the triangular fibrocartilage complex and undergoes arthroscopic repair
* Age between 19 and 60

Exclusion Criteria:

* Allergic to painkillers
* Have a serious heart rhythm
* epilepsy
* Severe pulmonary heart disease
* History of mental illness
* History of drug abuse
* received acupuncture treatment within 1 month

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
the effect of pain relief | in 36 hours after surgery
  Record the time required for the first injection of analgesics and the number of doses of oral painkiller and injection painkiller

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Cheng Chiu, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, No. 2, Yude Rd, North District, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No